CLINICAL TRIAL: NCT03688321
Title: Effects of Oral Probiotic Strains Lactobacillus Rhamnosus GR-1 and Lactobacillus Reuteri RC-14 on Prevention of GBS Vaginal Infection During Pregnancy and Influence of Postpartum Vaginal Health Condition.
Brief Title: Probiotic on Prevention of GBS Vaginal Infection During Pregnancy
Acronym: GBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMUH107-REC2-104
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Infection, Bacterial
Keywords: Probiotics; Group B Streptococcus; Infection; Prevention
MeSH Terms: conditions — Bacterial Infections; Infections | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Study Group: take 2 probiotics capsules before sleep for 12 weeks after being confirmed as GBS positive on 28th gestation Placebo Group: take 2 placebo capsules before sleep for 12 weeks after being confirmed as GBS positive on 28th gestation
Who Masked: Participant, Care Provider, Investigator
Masking Description: Labels with CMUH REC No. plus serial numbers on each bottle been completed by manufacturer and deliver to participants followed by random grouping order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic capsule GR-1 and RC-14 (Active Comparator): The intervention for study group is taking 2 capsules containing probiotic strains GR-1 and RC-14 before sleep for 18 weeks after being confirmed as GBS positive on 28th week gestation
  Interventions: Dietary Supplement: Probiotic capsule GR-1 and RC-14
- Placebo capsule (Placebo Comparator): The intervention for placebo group is taking 2 capsules not containing probiotic strains GR-1 and RC-14 before sleep for 18 weeks after being confirmed as GBS positive on 28th week gestation
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Probiotic capsule GR-1 and RC-14 — Study Group will take 2 probiotics capsules containing 1 billion colony forming unit(CFU) of Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 each before sleep for 18 weeks starting at 28th week gestation
  Other Names: U-relax
  Arms: Probiotic capsule GR-1 and RC-14
Dietary Supplement: Placebo capsule — Placebo Group will take 2 placebo capsules before sleep for 18 weeks starting at 28th week gestation
  Arms: Placebo capsule

SUMMARY:
The purpose of this study is to examine whether oral taking Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 from 28th week of gestation can reduce the GBS colonization rate of vagina and rectum in 35-37 weeks pregnant women as well as during laboring who present with GBS-positive at 28 weeks pregnancy. Through the results of our study, we try to investigate the role of probiotics in preventing the unnecessary tests, admission and antibiotic treatment in newborn with GBS-positive mother who deliver fewer than 4 hours after laboring and the influence of improving cervical diagnostics quality for postpartum Pap testing. Investigators hope the findings may have some effects on GBS sepsis and protocols as well as cervical diagnosis.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention(CDC) guideline in 2010 recommends minimum of 4 hours of intrapartum antibiotics prophylaxis on GBS colonized pregnant women for preventing early-onset GBS infection of neonates. However, GBS-positive mothers who arrive at the labor floor and deliver in fewer than 4 hours is frequent, especially in multiparous mothers. This problem is not easily resolved by antibiotic treatment of the pathogen; thus, such traditional approaches need to be reevaluated. The administration of specific Lactobacilli strains by mouth or intravaginally has been shown to be safe and effective in reducing urogenital infections. Previous results have showed that GR-1 and RC-14 can decrease GBS colonization during the later stage of pregnancy, taking probiotics capsules after GBS test in 35 to 37 weeks pregnant is still have to follow GBS guideline by CDC in 2010 of use antibiotics before delivery. Studies showed the use of antibiotics during pregnancy influenced the GI flora of neonates. Non-antibiotics prophylaxis for preventing newborns' GBS infection and reduce GBS colonization in 35-37 week pregnant are meaningful.

The raised estrogen and growth hormone during pregnancy may increase the activity of HPV molecule and human papilloma virus (HPV) infection. Short-time HPV persistence has been associated with higher risk for cervical intra-epithelial neoplasia and a higher risk of High-Grade Squamous Intraepithelial Lesion(HSIL). Clinical data showed GR-1 and RC-14 can improve the cervical malignancy diagnostics quality for non-pregnant women. The influence of oral probiotics on postpartum cervical diagnosis result is remain unknown.

This study is a prospective double blind randomized clinical trial. Vaginal and rectal GBS test are carried out at 28 weeks of gestation. Subjects with GBS-positive are invited to participate in this study after informed consent. 200 pregnant women are randomly assigned to one of the two groups. The study group is treated with two oral capsules of probiotics once daily (before sleeping) for 18 weeks, and the control group will take 2 capsules of placebos.

Vaginal and rectal GBS culture is repeated in 35-37 week of gestation and intrapartum period. All participators will treat according to GBS guideline by CDC in 2010. Cervical diagnosis will be completed at the 6th week after delivery. Through the results of this study, investigators try to investigate the role of probiotics in preventing the unnecessary tests, admission and antibiotic treatment in newborn with GBS positive mother who deliver fewer than 4 hours after laboring and the influence of improving cervical diagnostics quality for postpartum Pap testing. Investigators hope the findings may have some effects on GBS sepsis and protocols and cervical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years old pregnant women
* Singleton pregnancy
* GBS positive confirmed on 28th week gestation with informed consent form
* Agreed to abstain from the use of any systemic or intra-vaginal antibiotic, antifungal agents, or any other intravaginal product(e.g., contraceptive creams, lubricants, and douches) throughout the trial period.

Exclusion Criteria:

* Multiple gestations
* Impaired immunity, diabetes, or any other kind of significant disease or acute illness that could complicate the evaluation of the results
* Received vaginal or systemic antibiotics and antifungal therapy within 2 weeks of the screening visit
* Allergy or GI dysfunction history after taking probiotics or yogurt
* Constipation

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 204 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change of GBS result from positive to negative will be measured through GBS test for both vagina and rectum in 35-37 weeks pregnant women and during laboring. | 18 weeks
  100 participants with GBS positive result recruit on 28th week gestation for each group will recheck GBS colonization through GBS culture test of vagina and rectum in 35-37 weeks gestation as well as during laboring. The percentage of GBS positive turned to negative in the two time points will be measured for study group and placebo group.

SECONDARY OUTCOMES:
The number of normal, inflammation and atypical squamous cells(ASC-US) of the Papanicolaou Stain(PAP smear test) results for study group and placebo group will be measured through cervical PAP Smear Test on the 6th week after laboring. | 18 weeks
  100 participants of each group will be examined through cervical PAP smear test to collect the cases of participants with the result of normal, inflammation or ASC-US on the 6th week after laboring for cervical health condition analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ho, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical Univrsity Hoospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Ho M, Chang YY, Chang WC, Lin HC, Wang MH, Lin WC, Chiu TH. Oral Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 to reduce Group B Streptococcus colonization in pregnant women: A randomized controlled trial. Taiwan J Obstet Gynecol. 2016 Aug;55(4):515-8. doi: 10.1016/j.tjog.2016.06.003. PMID 27590374